CLINICAL TRIAL: NCT06074406
Title: Low-Field Bedside Magnetic Resonance Imaging for Detection of Acute Brain Injury in Pediatric Extracorporeal Membrane Oxygenation
Brief Title: Low-Field Bedside Brain Magnetic Resonance Imaging in Pediatric Extracorporeal Membrane Oxygenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Jessica S. Wallisch, Pediatric Intensivist, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY00002824
Record Dates: First submitted 2023-09-04; First posted 2023-10-10 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Feasibility and Safety of a Low-field MRI; Acute Brain Injury; Extracorporeal Membrane Oxygenation Complication
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Portable MRI Arm (Experimental): All subjects enrolled with be assigned to Arm 1
  Interventions: Device: Hyperfine

INTERVENTIONS:
Device: Hyperfine — Enrolled subjects will undergo a Hyperfine MRI exam, which is a portable, low-field MRI, at various timepoints during their clinical course on ECMO

SUMMARY:
The primary object of the study is to further characterize safety and feasibility of low-field bedside MRI in pediatric and neonatal ECMO patients. To perform imaging assessments of an early-stage magnetic resonance imaging (MRI) system on patients using low field magnetic strength. Collect qualitative data from the image assessments to optimize device performance using a low field magnetic resonance imaging device in a simulated use environment; Collect qualitative data from the image assessments using a high field magnetic resonance imaging, computed tomography and ultrasound devices. Generate anonymized image data for post-acquisition evaluation, performance measuring and planning for subsequent study size

ELIGIBILITY:
Inclusion Criteria

* Subjects admitted to the Pediatric Intensive Care Unit, Cardiac Intensive Care Unit, or the Neonatal Intensive Care Unit at Children's Mercy Kansas City
* Ages 0-17 years
* Undergoing venovenous or venoarterial ECMO

Exclusion Criteria

* Pregnancy
* Active implants such as:

  * Pacemaker
  * Implanted defibrillator
  * Implanted insulin pump
  * Deep brain stimulator
  * Vagus nerve stimulator
  * Cochlear implant
  * Programmable shunt
* MRI incompatible surgical hardware (e.g., staples, screws, etc.)
* Metal-containing tattoos or permanent make-up on head or neck
* Suspected metal in eye, e.g.,
* Former or current welders, metal workers, or individuals with a metal injury
* Metal shrapnel
* Passive implants are considered MRI conditional

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Examining the occurrence of adverse events and serious adverse events with portable MRI use in ECMO patients | During Intervention, and immediately after intervention.
  Measuring the occurrence of adverse events and serious adverse events that occurring during the portable MRI procedure. Adverse events and serious adverse events include (change in mean arterial pressure by 20% increase or decreased measured by the meters of mercury as identified by catheter measurement in patient, a decrease in the ECMO flow rate by 20% measured in milliliters per min by the ECMO machine, decrease in the oxygen saturation by 10% measured by pulse oximetry, dislodgement of the ECMO cannula measured by the occurrence of hemorrhage, as identified by PI).
Assessing the time needed to conduct a portable MRI with ECMO patients. | Pre intervention during patient prep, and during intervention, and immediately intervention.
  The analyses will examine the amount of time it takes to conduct a Portable MRI with ECMO patients. The examination records the amount of time to prep and move the patient to the portable MRI and back from the portable MRI. Preparation and movement of patient will be measured using a stopwatch identifying the number of minuets passed. The amount of time it takes to conduct the portable MRI with ECMO patients will also be analyzed. The time the MRI takes will be measured using a stopwatch examining the number of minuets passed.
Analyzing the number of staff required to conduct a Portable MRI with an ECMO patient. | Pre intervention, during intervention, and immediately after intervention.
  The analysis will examine the number of staff needed to prep and use a portable MRI with patients. Number of staff needed will be record in RedCap via head count.
Determine the number of critical care therapies conducted during imaging studies. | Pre intervention during patient prep, during intervention, and immediately after intervention.
  Analyzing the number of critical therapies conducted during patient prep, during intervention, and post intervention. The study will record in RedCap the number of critical care therapies identified by study coordinator and PI by counting the number of therapies. Critical care therapies include (EEG, mechanical ventilation, continuous renal replacement therapy, continuous IV infusions, temporary pacing wires).

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Wallisch, MD, Principal Investigator — Children's Mercy Kansas City
Locations (1):
- Children's Mercy Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wallisch JS, Wagner AF, Daniel JM, Taber A, Sien M, Foster S, Artz N, Zinkus TP, Yeh HW, Pineda JA, Kochanek PM, Chan SS. Ultra-Low-Field Portable Magnetic Resonance Imaging Feasibility and Safety in Pediatric and Neonatal Extracorporeal Membrane Oxygenation: A Single-Center Year-Long Experience. J Am Heart Assoc. 2025 Nov 18;14(22):e043434. doi: 10.1161/JAHA.125.043434. Epub 2025 Nov 11. PMID 41220148